CLINICAL TRIAL: NCT01344668
Title: The Public Private Partnership Addressing Literacy-Numeracy to Improve Diabetes Care
Acronym: PRIDE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Russell Rothman, Principal Investigator, Vanderbilt University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 101523; 1R18DK083264-01A2 (NIH)
Record Dates: First submitted 2011-04-27; First posted 2011-04-29 (Estimated); Last update posted 2016-10-14 (Estimated); Status verified 2016-10

CONDITIONS: Type 2 Diabetes
Keywords: Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard Diabetes Education (Other): Standard Diabetes Education
  Interventions: Other: Standard Diabetes Education
- Enhanced Diabetes Education (Other): Enhanced Diabetes Education
  Interventions: Other: Enhanced Diabetes Education

INTERVENTIONS:
Other: Enhanced Diabetes Education — Provide enhanced diabetes education
  Arms: Enhanced Diabetes Education
Other: Standard Diabetes Education — Provide Standard Diabetes Education
  Arms: Standard Diabetes Education

SUMMARY:
The primary hypotheses are that the intervention will improve A1C, blood pressure, lipids, weight, self-efficacy, self-management behaviors, and use of clinical services at 12 and 24 months follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Patient has a clinical diagnosis of Type 2 Diabetes
* Age 18-85 years
* English or Spanish speaking
* Most recent A1C ≥ 7.5%
* Patient agrees to participate in the study for the full two years duration.

Exclusion Criteria:

* Poor visual acuity (vision worse than 20/50 using Rosenbaum Pocket Screener) -- Significant dementia or psychosis (by health provider report or chart review)
* Terminal illness with anticipated life expectancy < 2 years (per health provider or patient report).

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 411 (Actual)
Dates: Start 2011-05; Primary Completion 2015-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Improvement in A1C at 12 months | 12 months
  The primary outcome will be the improvement in A1C at 12 months between Intervention group patients and Control group patients.

CONTACTS AND LOCATIONS:
Overall Officials: Russell L. Rothman, MD, MPP, Principal Investigator — Vanderbilt University
Locations (1):
- Vanderbilt University, Nashville, Tennessee, United States